CLINICAL TRIAL: NCT03472716
Title: The βIG-H3 Protein: a New Marker in PANCreatic Adenocarcinoma
Brief Title: The βIG-H3 Protein: a New Marker in PANCreatic Adenocarcinoma (BIGHPANC)
Acronym: BIGHPANC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: BIGHPANC - ET17-113
Record Dates: First submitted 2018-02-27; First posted 2018-03-21 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Pancreas Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; βig-h3; Pronostic marker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (included in the standard care) at inclusion and in case of relapse.
  Initial tumoral sample from the surgical exeresis or from the sample obtained for the initial diagnosis (metastases biopsies) and new tumoural sample in case of relapse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Samples: Included patients will undergo 2 biological samples : a 5-ml blood sample included in the standard care and a tumoral sample (from the surgical exeresis or from the initial diagnosis biopsy). Patients with a confirmed pancreatic carcinoma will be followed during 18 months in this cohort. In case of relapse, patients will have 2 new biological samples (blood and tumoral).
  Interventions: Procedure: Biological Samples

INTERVENTIONS:
Procedure: Biological Samples — 5 ml blood sample and one tumoural sample (either a fresh biopsy or the initial diagnosis biopsy).
  In case of relapse, new samples will be performed (blood and tumoral samples)

SUMMARY:
The primary objective of this trial is to evaluate the correlation between the intensity of the protein big-h3 expression at tumoural microenvironment and the TNM/UICC staging (from I to IV) of pancreatic adenocarcinoma lesion.

DETAILED DESCRIPTION:
The pancreatic adenocarcinoma is the most common pancreatic cancer. Currently, it represents the fourth cause of death by cancer in France. The diagnosis is often realized when the disease is at an advanced stage because of its delayed clinical expression. Only 20% of the patients are diagnosed at a stage enabling a tumour resection.

Scientists discovered a protein playing a key role: the βig-h3 protein. In mouse models, this protein is present in several stages of the tumorigenesis. A mutation of the gene Kras leads to the development of PANin (Pancreatic Intraepithelial Neoplasia) type precancerous lesions. The βig-h3 protein is early and highly expressed in the stroma around these lesions and in the pancreatic adenocarcinoma stroma. Moreover, studies showed that protein neutralization leads to a tumour size reduction by increasing the CD8+anti-tumor activity.

This protein is detected in the blood serum of patients suffering from a pancreatic adenocarcinoma. So, this protein which is secreted by the extracellular matrix could be a predictive marker for the pancreatic adenocarcinoma.

In this prospective, multicentric non-interventional study, it is anticipated to recruit 80 patients (20 per TNM/UICC stage).

Included patients will undergo two samples: A blood sample (5 ml) and a tumour sample (surgical exeresis piece or tumour tissue obtained for the initial diagnosis). In case of relapse, new samples will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the day of consenting to the study
* Patient with a potential pancreatic adenocarcinoma whatever the TNM/UICC stage
* Systematic treatment not initiated
* Signed and dated informed consent document.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Geographical, social or psychiatric reason preventing the patient from completing the study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting a pancreatic adenocarcinoma (TNM/UICC from I to IV) having given a written consent for participating to the study. Patients are to be followed up until the LVLP (minimum duration: 18 months, maximum: 36 months)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the correlation between the intensity of the protein βig-h3 expression at tumoural microenvironment and the TNM/UICC (from I to IV) of pancreatic adenocarcinoma lesion | At inclusion
  Correlation between the intensity of the protein βig-h3 expression at tumoural microenvironment and the TNM/UICC (from I to IV) of pancreatic adenocarcinoma lesionimmunohistochemical analysis of pancreatic adenocarcinoma

SECONDARY OUTCOMES:
Evaluation of the correlation of βig-h3 protein blood rate and the pancreatic adenocarcinoma TNM/UICC staging | At inclusion and upon relpase assessed up to 36 months
  Correlation between βig-h3 protein blood rate (ELISA) and the pancreatic adenocarcinoma TNM/UICC staging
Evaluation of the correlation between the βig-h3 protein expression intensity in the tumoural microenvironment and the immune infiltrate LT CD8+ of pancreatic adenocarcinoma | At inclusion and upon relpase assessed up to 36 months
  Correlation between the βig-h3 protein expression intensity in the tumoural microenvironment and the immune infiltrate LT CD8+ of pancreatic adenocarcinoma
Evaluation of the correlation between βig-h3 protein expression intensity and patients clinical evolution | 6 months after patient's inclusion
  Correlation between βig-h3 protein expression intensity and patients clinical evolution (6-month objective response rate according to RECIST 1.1 criteria)
Evaluation of the the correlation between βig-h3 protein expression intensity and patients clinical evolution | Assessed up to 36 months
  Correlation between βig-h3 protein expression intensity and Overall Survival
Evaluation of the correlation between βig-h3 protein expression intensity and patients clinical evolution | Assessed up to 36 months
  Correlation between βig-h3 protein expression intensity and Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: DE LA FOUCHARDIERE Christelle, Dr, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France